CLINICAL TRIAL: NCT05219019
Title: Feasibility of Remote Measures and Assessments in Deep Brain Stimulation for Parkinson's Disease (FoRMA-DBS)
Acronym: FoRMA-DBS
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient interest by potential participants.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: H-41349
Record Dates: First submitted 2021-12-14; First posted 2022-02-01 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
Keywords: Deep brain stimulation (DBS); Remote monitoring; Subthalamic nucleus (STN); Internal globus pallidus (GPi); Patient Global Impression of Change (PGIC); Activities Balance Confidence Scale (ABC); Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD patients who have elected DBS: Ten individuals with moderate to advanced Parkinson's disease who have elected to undergo deep brain stimulation (DBS) of the subthalamic nucleus (STN) or internal globus pallidus (GPi) as standard of care for management of Parkinson's disease tremor and/or motor complications

SUMMARY:
This is an observational pilot study to assess the feasibility of remote functional assessments of gait, balance, and functional mobility via a telemedicine platform enabled via the Abbott Infinity devices. The clinical care of the participant will not be changed based on the remote functional assessments.

DETAILED DESCRIPTION:
This is a single-center, non-randomized pilot observational study to explore the feasibility and tolerability of remotely assessing gait speed, functional mobility and balance measures in patients with Parkinson's disease experiencing medication-refractory tremor, motor complications and/or dyskinesias undergoing initiation of deep brain stimulation therapy. This study explores the feasibility of remotely performing and collecting functional assessments of gait, balance and mobility in the setting of programming deep brain stimulation (DBS).

Ten participants who are deemed surgical candidates for receiving DBS for Parkinson's disease under standard of clinical care processes (neuropsychological testing, neurology consultation and neurosurgery consultation) and have opted for the Abbott DBS system will be enrolled in the study and undergo the pre-surgical and post-surgical visits. A pre-operative in-clinic visit will take place approximately 28 days (day -42) prior to surgical DBS electrode lead implantation. An at-home assessment will take place within 14 days (day -28) of this baseline visit, still prior to surgical DBS electrode lead implantation. Participants will receive care as usual including their first post-operative clinic visit for initial programming (day 28), just like standard of care for DBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with with Parkinson's disease, as confirmed by the treating investigator, providing written consent to the clinical study
* Participants have been determined by the treating investigator as candidates for DBS
* Participants who have opted to have DBS with the remote-programming capable platform
* Have internet connection at home or wherever participants will be receiving care remotely and be able to participate in telemedicine visits and remote programming

Exclusion Criteria:

* Has already had prior surgical lesioning or deep brain stimulation therapy
* Meets criteria for Parkinson's disease dementia in the opinion of the treating investigator
* Does not have capacity for consent as judged by the treating investigator
* Scores less than 24 on the Montreal Cognitive Assessment (MoCA) at standard of care DBS screening, indicating, at least, mild cognitive impairment

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with moderate to advanced Parkinson's disease who have elected to undergo deep brain stimulation (DBS) of the subthalamic nucleus (STN) or internal globus pallidus (GPi) as standard of care for management of Parkinson's disease tremor and/or motor complications
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of remotely assessing gait speed during DBS therapy initiation | 20 weeks
  A telemedicine platform enabled via the Abbott Infinity device will be used to remotely assess gait speed.
Feasibility of remotely assessing functional mobility during DBS therapy initiation | 20 weeks
  A telemedicine platform enabled via the Abbott Infinity device will be used to remotely assess functional mobility.
Feasibility of remotely assessing balance during DBS therapy initiation | 20 weeks
  A telemedicine platform enabled via the Abbott Infinity device will be used to remotely assess balance.

SECONDARY OUTCOMES:
Mobility assessment: 4 meter walk | days -42, -28, 21, 28, 42, 56, 70, and 84
  Gait speed as performed during the 4-meter walk: Measured as time taken to walk 4 meters in seconds.
Mobility assessment: Timed up and go (TUG) | days -42, -28, 21, 28, 42, 56, 70, and 84
  The TUG assesses mobility, balance, walking ability and fall risk in older adults and has been validated showing good agreement between in-person and telehealth and raters. On the command, "go" the patient rises from the chair, walks 3 meters at a comfortable safe pace, turns and walks back to the chair and sits down. Measured as time taken to complete task in seconds.
Mobility assessment: 5 times sit to stand | days -42, -28, 21, 28, 42, 56, 70, and 84
  This is a timed task that requires the participant to stand from a seated position five times in a row. Measured as time taken to complete task in seconds.
Mobility assessment: 360 degree turns | days -42, -28, 21, 28, 42, 56, 70, and 84
  The 360 degree turn test is a measure of dynamic balance in which the participant turns in a complete circle. Measured as time taken to complete task in seconds.
Mobility assessment: Activity-specific balance confidence (ABC) scale | days -42, -28, 21, 28, 42, 56, 70, and 84
  Self-reported confidence in performing 16 activities without losing balance. Participants rate using an 11-point likert-type scale, from 0% (no confidence) to 100% (completely confident) with 10% increments. A total score will be calculated as the mean of the items.
Mobility assessment: Single-leg stance | Day -28, 21, 42, 56, 70
  Amount of time participant is able to stand on one leg (performed for each leg), measured in seconds.
Movement disorders | day -42 and day 84
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I-IV
  The Movement Disorder Society's Unified Parkinson's Disease Rating Scales (MDS-UPDRS) consists of 65 items across four domains: non-motor experiences, motor experiences, a motor examination, and motor complications, rated from 0 (normal) to 4 (severe). Subscales and a total score are calculated by adding items. A higher score is a worse outcome and indicates more severe symptoms of Parkinson's disease.
Quality of Life in PD | day -42 and day 84
  The Parkinson's Disease Questionnaire (PDQ-39) will be used to assess living difficulties across 8 dimensions of daily living including mobility subscores.
  The PDQ-39 assesses life concerns of individuals with PD. It is composed of a summary index and eight domain scores-mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. Each item is rated on a 0 (never) to 4 (always) scale. A higher score indicates a higher self-perceived frequency of quality of life and health problems in the past month that are due to the disease, with each domain normed to a scale on which 0 indicating never a problem and 100 always a problem. The summary index is the average of the normed domain scores. A higher score is a worse outcome for quality of life.
Change in 3-day step count before DBS | day -42, day 84
  Step count will be measured continuously by a StepWatch4 over a 3 day period.
Change in amount of time spent with tremor and dyskinesia | baseline, day 84
  The amount of time spent with tremor and dyskinesia will be measured with the Apple watch.
Patient global impression of change | baseline, day 28, 42, 56, 70 and 84
  The Patient Global Impression - Improvement scale (CGI-I) is a 7 point scale, from 1 (normal) through to 7 (amongst the most severely ill), that requires the patient to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the study. Higher scores reflect more severe illness.
Clinician global impression of change | baseline, day 28, 42, 56, 70 and 84
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale, from 1 (normal) through to 7 (amongst the most severely ill), that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the study. Higher scores reflect more severe illness.

CONTACTS AND LOCATIONS:
Overall Officials: Ludy Shih, MD MMSc, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck CA, Beran DB, Biglan KM, Boyd CM, Dorsey ER, Schmidt PN, Simone R, Willis AW, Galifianakis NB, Katz M, Tanner CM, Dodenhoff K, Aldred J, Carter J, Fraser A, Jimenez-Shahed J, Hunter C, Spindler M, Reichwein S, Mari Z, Dunlop B, Morgan JC, McLane D, Hickey P, Gauger L, Richard IH, Mejia NI, Bwala G, Nance M, Shih LC, Singer C, Vargas-Parra S, Zadikoff C, Okon N, Feigin A, Ayan J, Vaughan C, Pahwa R, Dhall R, Hassan A, DeMello S, Riggare SS, Wicks P, Achey MA, Elson MJ, Goldenthal S, Keenan HT, Korn R, Schwarz H, Sharma S, Stevenson EA, Zhu W; Connect.Parkinson Investigators. National randomized controlled trial of virtual house calls for Parkinson disease. Neurology. 2017 Sep 12;89(11):1152-1161. doi: 10.1212/WNL.0000000000004357. Epub 2017 Aug 16. PMID 28814455
- [Background] Collomb-Clerc A, Welter ML. Effects of deep brain stimulation on balance and gait in patients with Parkinson's disease: A systematic neurophysiological review. Neurophysiol Clin. 2015 Nov;45(4-5):371-88. doi: 10.1016/j.neucli.2015.07.001. Epub 2015 Aug 28. PMID 26319759
- [Background] Deuschl G, Schade-Brittinger C, Krack P, Volkmann J, Schafer H, Botzel K, Daniels C, Deutschlander A, Dillmann U, Eisner W, Gruber D, Hamel W, Herzog J, Hilker R, Klebe S, Kloss M, Koy J, Krause M, Kupsch A, Lorenz D, Lorenzl S, Mehdorn HM, Moringlane JR, Oertel W, Pinsker MO, Reichmann H, Reuss A, Schneider GH, Schnitzler A, Steude U, Sturm V, Timmermann L, Tronnier V, Trottenberg T, Wojtecki L, Wolf E, Poewe W, Voges J; German Parkinson Study Group, Neurostimulation Section. A randomized trial of deep-brain stimulation for Parkinson's disease. N Engl J Med. 2006 Aug 31;355(9):896-908. doi: 10.1056/NEJMoa060281. PMID 16943402
- [Background] Dorsey ER, Achey MA, Beck CA, Beran DB, Biglan KM, Boyd CM, Schmidt PN, Simone R, Willis AW, Galifianakis NB, Katz M, Tanner CM, Dodenhoff K, Ziman N, Aldred J, Carter J, Jimenez-Shahed J, Hunter C, Spindler M, Mari Z, Morgan JC, McLane D, Hickey P, Gauger L, Richard IH, Bull MT, Mejia NI, Bwala G, Nance M, Shih L, Anderson L, Singer C, Zadikoff C, Okon N, Feigin A, Ayan J, Vaughan C, Pahwa R, Cooper J, Webb S, Dhall R, Hassan A, Weis D, DeMello S, Riggare SS, Wicks P, Smith J, Keenan HT, Korn R, Schwarz H, Sharma S, Stevenson EA, Zhu W. National Randomized Controlled Trial of Virtual House Calls for People with Parkinson's Disease: Interest and Barriers. Telemed J E Health. 2016 Jul;22(7):590-8. doi: 10.1089/tmj.2015.0191. Epub 2016 Feb 17. PMID 26886406
- [Background] GBD 2016 Parkinson's Disease Collaborators. Global, regional, and national burden of Parkinson's disease, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):939-953. doi: 10.1016/S1474-4422(18)30295-3. Epub 2018 Oct 1. PMID 30287051
- [Background] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Background] Li D, Zhang C, Gault J, Wang W, Liu J, Shao M, Zhao Y, Zeljic K, Gao G, Sun B. Remotely Programmed Deep Brain Stimulation of the Bilateral Subthalamic Nucleus for the Treatment of Primary Parkinson Disease: A Randomized Controlled Trial Investigating the Safety and Efficacy of a Novel Deep Brain Stimulation System. Stereotact Funct Neurosurg. 2017;95(3):174-182. doi: 10.1159/000475765. Epub 2017 Jun 2. PMID 28571034
- [Background] Ma Y, Miao S, Zhou R, Zhang Q, Chen H, Liang Y. Application of Remote Deep Brain Stimulation Programming for Parkinson's Disease Patients. World Neurosurg. 2021 Mar;147:e255-e261. doi: 10.1016/j.wneu.2020.12.030. Epub 2020 Dec 13. PMID 33316487
- [Background] Powers R, Etezadi-Amoli M, Arnold EM, Kianian S, Mance I, Gibiansky M, Trietsch D, Alvarado AS, Kretlow JD, Herrington TM, Brillman S, Huang N, Lin PT, Pham HA, Ullal AV. Smartwatch inertial sensors continuously monitor real-world motor fluctuations in Parkinson's disease. Sci Transl Med. 2021 Feb 3;13(579):eabd7865. doi: 10.1126/scitranslmed.abd7865. PMID 33536284
- [Background] Schuepbach WM, Rau J, Knudsen K, Volkmann J, Krack P, Timmermann L, Halbig TD, Hesekamp H, Navarro SM, Meier N, Falk D, Mehdorn M, Paschen S, Maarouf M, Barbe MT, Fink GR, Kupsch A, Gruber D, Schneider GH, Seigneuret E, Kistner A, Chaynes P, Ory-Magne F, Brefel Courbon C, Vesper J, Schnitzler A, Wojtecki L, Houeto JL, Bataille B, Maltete D, Damier P, Raoul S, Sixel-Doering F, Hellwig D, Gharabaghi A, Kruger R, Pinsker MO, Amtage F, Regis JM, Witjas T, Thobois S, Mertens P, Kloss M, Hartmann A, Oertel WH, Post B, Speelman H, Agid Y, Schade-Brittinger C, Deuschl G; EARLYSTIM Study Group. Neurostimulation for Parkinson's disease with early motor complications. N Engl J Med. 2013 Feb 14;368(7):610-22. doi: 10.1056/NEJMoa1205158. PMID 23406026
- [Background] Soileau MJ, Persad C, Taylor J, Patil PG, Chou KL. Caregiver burden in patients with Parkinson disease undergoing deep brain stimulation: an exploratory analysis. J Parkinsons Dis. 2014;4(3):517-21. doi: 10.3233/JPD-140380. PMID 24903924
- [Background] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Background] Xu J, Wang J, Keith S, Zhang M, Yang C, Yuan Q, Qiu Y, Hu X, Wu X. Management of Parkinson's disease patients after DBS by remote programming: preliminary application of single center during quarantine of 2019-nCoV. J Neurol. 2021 Apr;268(4):1295-1303. doi: 10.1007/s00415-020-10273-z. Epub 2020 Oct 26. PMID 33104873
- [Background] Chen Y, Hao H, Chen H, Li L. The study on a telemedicine interaction mode for Deep Brain Stimulation postoperative follow-up. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:186-9. doi: 10.1109/EMBC.2015.7318331. PMID 26736231
- [Background] Zhang C, Zhu K, Lin Z, Huang P, Pan Y, Sun B, Li D. Utility of Deep Brain Stimulation Telemedicine for Patients With Movement Disorders During the COVID-19 Outbreak in China. Neuromodulation. 2021 Feb;24(2):337-342. doi: 10.1111/ner.13274. Epub 2020 Oct 2. PMID 33006811
- [Background] Zhang J, Hu W, Chen H, Meng F, Li L, Okun MS. Implementation of a Novel Bluetooth Technology for Remote Deep Brain Stimulation Programming: The Pre- and Post-COVID-19 Beijing Experience. Mov Disord. 2020 Jun;35(6):909-910. doi: 10.1002/mds.28098. Epub 2020 Jun 1. No abstract available. PMID 32478886